CLINICAL TRIAL: NCT02764723
Title: Isobaric Ropivacaine 15 mg Versus Hyperbaric Bupivacaine 12.5 mg for Spinal Anesthesia in Geriatric Patients Undergoing Total Knee Arthroplasty
Brief Title: Isobaric Spinal Ropivacaine Versus Hyperbaric Spinal Bupivacaine in Total Knee Arthroplasty in Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Sayed Mohamed Abbas (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sayed Mohamed Abbas, Doctor, Al Mouwasat Hospital
Organization: Al Mouwasat Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSAT-3
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Total Knee Arthroplasty in Geriatric Patients; Spinal Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyperbaric bupivacaine (Active Comparator): 12.5 mg of 0.5% hyperbaric bupivacaine
  Interventions: Drug: Hyperbaric bupivacaine
- Isobaric ropivacaine (Experimental): 15 mg of 0.5% isobaric ropivacaine
  Interventions: Drug: Isobaric ropivacaine

INTERVENTIONS:
Drug: Hyperbaric bupivacaine — 12.5 mg of hyperbaric bupivacaine 0.5% for spinal anesthesia in geriatric patients undergoing total knee arthroplasty
  Arms: Hyperbaric bupivacaine
Drug: Isobaric ropivacaine — 15 mg of isobaric ropivacaine 0.5% for spinal anesthesia in geriatric patients undergoing total knee arthroplasty
  Arms: Isobaric ropivacaine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of spinal anesthesia with isobaric ropivacaine, compared with hyperbaric bupivacaine in geriatric patients undergoing lower limb orthopedic surgery.

DETAILED DESCRIPTION:
52 patients physical status II-III according to the American Society of Anesthesiologists classification aged 65 years and above of average height, and scheduled for total knee replacement under spinal anesthesia.

Patients were randomly assigned into two equal groups of 26 patients each according to the type of local anesthetic injected in the subarachnoid space , Group I : patients who received an intrathecal injection of 12.5 mg of 0.5% hyperbaric bupivacaine , Group II: patients who received an intrathecal injection of 15 mg of 0.5% ropivacaine.

The investigators compared both groups as regards the extent and duration of sensory and motor block and hemodynamics including heart rate (HR) , non invasive mean arterial blood pressure (MAP) and respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status II-III aged 65 years and above of average height, and scheduled for total knee replacement under spinal anesthesia.

Exclusion Criteria:

* Known hypersensitivity to amide local anesthetics and contraindications to spinal anesthesia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in the extent and duration of sensory block | within 2 years
  The assessment of sensory block to pinprick was performed at 2, 4, 6, 8, 10, and 15 min after the intrathecal injection and then every 15 min until regression to L5. Results of the pinprick test were determined bilaterally at midclavicular level by using a short-beveled 27-gauge needle. Response to pain we determined by asking the patient whether or not he feels pain with the pinprick.
Changes in the extent and duration of motor block | within 2 years
  Motor block in the lower limb was assessed by using a modified Bromage scale (0 = no paralysis , 1 = unable to raise extended leg , 2 = unable to flex knee , 3 = unable to flex ankle). These assessments were performed immediately after the assessments of sensory block until the return of normal motor function.
Changes in the heart rate | within 2 years
  All patients of these 2 groups were assessed and monitored for Haemodynamics using ECG for heart rate (HR). Baseline values were defined as heart rate values before the preanesthetic infusion. The values were recorded before the induction and then every 5 min until discharge from the recovery room.
Changes in the non invasive mean arterial blood pressure | within 2 years
  All patients of these 2 groups were assessed and monitored for Haemodynamics as regards non invasive mean arterial blood pressure (MAP). Baseline values were defined as blood pressure values before the preanesthetic infusion. The values were recorded before the induction and then every 5 min until discharge from the recovery room.
Respiratory depression | within 2 years
  Respiratory depression (defined as respiratory rate < 8 min and SPO 2 < 90%)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] D'Souza AD, Saldanha NM, Monteiro AD. Comparison of Intrathecal Hyperbaric 0.5% Bupivacaine, Isobaric 0.5% Levobupivacaine and Isobaric 0.75% Ropivacaine for Lower Abdominal Surgeries. International Journal of Health Sciences and Research (IJHSR). 2014;4(1):22-9.